CLINICAL TRIAL: NCT06771804
Title: Cricket Flour Metabolism in Humans
Acronym: InsectGEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FHMS 21-22 231 EGA
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Nutrition, Healthy
Keywords: Nutrition; Alternative Protein; Gastric emptying
MeSH Terms: interventions — capsid protein, Cricket paralysis virus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Whey Protein intervention
  Interventions: Dietary Supplement: Cricket Protein
- Insect (Experimental): Cricket Protein intervention
  Interventions: Dietary Supplement: Cricket Protein

INTERVENTIONS:
Dietary Supplement: Cricket Protein — Participants are provided with muffins containing either whey or cricket protein.

SUMMARY:
With increasing demands on the environment people are looking in different ways to decrease their carbon footprint. Protein is an important part of human diets a it provides building blocks for growth and helps to ensure people stay health. Animal protein is one of the primary sources of of protein from our diets but it is also known that farming cattle for example places a lot of pressure on the environment. As a result of this new protein sources are being looked at that can take the place of animal protein. Insects have been consumed on many civilisations for a long time and they are slowly making their way into the western diets.

At this time the investigators however do not know very much about how well insect protein compares to animal protein as a nutritious food source. This research project is therefore one of the first to compare some of the nutritional properties between animal and insect proteins.

In brief, this study involves eating a sweet breakfast muffin made of either whey (animal) protein powder or cricket flour (very finely ground whole adult crickets) and then breathing into test tubes at various time points for a few hours as well as collecting some small amounts of blood using a finger stick to measure blood glucose and fats.

DETAILED DESCRIPTION:
Insects have been used as protein source for many years in East-Asian and African populations, and more recently the interest in this potential protein source has been growing in Western countries due to the issues outlined above and increased awareness of animal welfare issues in the food chain. However, up until now there is no clear evidence that insect-derived protein has the same nutritional properties as its animal counterpart. Even though nutritional composition of insects can be similar or sometimes even better to support a healthy diet certain properties of the insects (such as the chitin in their exoskeleton) could have detrimental effects on their bioavailability. Gastric emptying (GE) describes the process of food being digested and absorbed by the controlled delivery from the stomach into the duodenum (1.). In the field of nutrition, GE is important, since a slower rate of GE can lead to a lower postprandial rise in macronutrients, and consequently a lower postprandial burden on their clearance. To date it is known that certain food properties such as volume, calories, and viscosity, as well as physiological factors such as age and gender can influence the gastric emptying rate (1.). However, the interaction between human physiology and different food in the stomach is widely unknown.

A slower GE rate is particularly important regarding postprandial plasma triacylglycerol concentrations, with impaired clearance being related to inflammation and cardiovascular disease. The attenuation of the postprandial increase in blood glucose has long been a goal for improved metabolic health. As reviewed, small differences in GE can have a major impact on postprandial glycaemia in health and type 2 diabetes (2.). Furthermore, a slowed gastric emptying rate as a result of certain types of food is associated with a delayed reoccurrence of feeling of hunger and can influence satiation.

The 13C octanoic acid breath test is a relatively cheap, non-invasive, and simple test to measure GE. The test is performed via the ingestion of a controlled meal containing the commercially available non-harmful stable isotope 13C in a short chain fatty acid (C8) and the following detection of the 13Clabelled CO2 in the breath (3.).

The data generated by the breath test is commonly analysed with a one compartment model based on Ghoos et al (1993) (4.) to generate parameters such as half time and lag time. More advanced semi mechanistic models are used in pharmacokinetics and could be applied to the breath test.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adult males and females between 20 and 55 years of age

  * BMI between 18.5 and 35 kg/m2
  * Weight stable for 3 months (± 2 kg)
  * Volunteers must be able and willing to give informed written consent
  * Volunteers must be able to eat egg (because egg is required for preparation of the stable isotope dosage see section experimental design).

Exclusion Criteria:

* Previous or current medical conditions, including heart disease, diabetes, gastrointestinal diseases (for example Crohn's disease, Coeliac disease, Inflammatory Bowel Disease), liver disease, endocrine diseases - assessed via a health questionnaire (appendix)
* Those taking (or have been taking within the past 6 months) regular medication, excluding contraceptive medication, or food supplements (e.g., vitamins, minerals, fish oil, fibre supplements, antioxidant tablets) - assessed via a health questionnaire (appendix) Those smoking, using nicotine products (e.g., e-cigarettes, patches) or not abstained from these activities for more than 6 months
* Pregnant or lactating
* Volunteers with a habitual caffeine intake > 300 mg/day (more than 5 cups standard coffee)
* Drug or alcohol abuse in the last 2 years
* The principal investigator considers it unsafe / unsuitable for the volunteer to be in the study
* Those who are currently taking part in a clinical trial or another research study or have taken part within the last 3 months
* Those who do not refrain from alcohol, caffeine containing drinks (e.g., coffee, coca cola, tea, Red Bull) and strenuous exercise 10 hours before the laboratory session
* Those with food allergies, dietary intolerance (especially for egg), or Coeliac disease
* Those following weight reducing diets

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Digestion | 4 hours post prandial
  Gastric emptying

SECONDARY OUTCOMES:
Digestion | 4 hours post prandial
  T lag
Blood metabolites | 4 hours post prandial
  Glucose
Blood metabolites | 4 hours post prandial
  Cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD is planned